CLINICAL TRIAL: NCT00861016
Title: An Open-Label, Non-Comparative, Multi-Centre Study to Evaluate the Efficacy and Safety of Metoprolol Succinate Prolonged-Release Tablet (Betaloc Zok) in Patients With Mild to Moderate Essential Hypertension
Brief Title: Efficacy and Safety of Metoprolol Succinate Prolonged-Release Tablet in Patients With Mild to Moderate Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Marco Avila, AstraZeneca Pharmaceuticals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D4025L00006
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-03-13 (Estimated); Status verified 2009-03

CONDITIONS: Hypertension
Keywords: Post marketing study
MeSH Terms: conditions — Hypertension | interventions — Felodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): The patients with mild to moderate essential hypertension
  Interventions: Drug: metoprolol succinate prolonged-release tablet and felodipine

INTERVENTIONS:
Drug: metoprolol succinate prolonged-release tablet and felodipine — a regimen that starts with metoprolol succinate prolonged-release tablet 47.5mg once daily, orally and allows for dose escalation to 95mg once daily, orally at 4 weeks if not controlled; at week 8 allows for the addition of felodipine sustained release tablet 5mg once daily, orally
  Other Names: Betaloc ZOK and Plendil

SUMMARY:
This is an open-label, non-comparative, multi-centre clinical study to evaluate the Efficacy and safety of Metoprolol Succinate prolonged-release tablet (Betaloc Zok) in patients with mild to moderate essential hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Newly diagnosed essential hypertension who have not received anti- hypertensive treatment, or patients without antihypertensive medication in two weeks before screening, 90mmHg<SiDBP <110mmHg and SiSBP <180mmHg.

Exclusion Criteria:

* Known or suspected secondary hypertension
* Resting HR is < 55bpm.
* Sick sinus syndrome
* Atrioventricular block of first degree (with P-R>0.24seconds), or second or third degree

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2005-10; Primary Completion 2006-04 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Percent of subjects reaching blood pressure target at wk 8 after metoprolol succinate prolonged release tablet treatment, and magnitude of systolic and diastolic blood pressure reduction from baseline among subjects who reached target (below 140/90mmHg). | Day -7- -1, Day1, Day 28, Day 56,Day 84

SECONDARY OUTCOMES:
The magnitude of systolic and diastolic blood pressure reduction from baseline among all the subjects at week 8 after metoprolol succinate prolonged release tablet treatment. | Day -7- -1, Day1, Day 28, Day 56,Day 84
The percentage of subjects reaching blood pressure target at week 4, and the magnitude of systolic and diastolic blood pressure reduction from baseline among all the subjects and those subjects who reached target | Day -7- -1, Day1, Day 28, Day 56,Day 84
The percentage of subjects reaching blood pressure target at week 12, and the magnitude of systolic and diastolic blood pressure reduction from baseline among all the subjects and those subjects who reached target | Day -7- -1, Day1, Day 28, Day 56,Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Lisheng Liu, Principal Investigator — BeiJing Hypertension League